CLINICAL TRIAL: NCT01351649
Title: Middle School Physical Activity Intervention for Girls
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Lorraine Robbins, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HL090705 (NIH)
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Physical Activity
Keywords: exercise; adolescent; intervention; female; counseling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- attention control (Other): Sessions with school nurse to discuss health-promoting topics and after-school health-promoting workshop. Physical activity and healthy eating were not addressed.
  Interventions: Behavioral: middle school physical activity intervention for girls
- physical activity (Experimental)
  Interventions: Behavioral: middle school physical activity intervention for girls

INTERVENTIONS:
Behavioral: middle school physical activity intervention for girls — Both the "Girls on the Move" intervention and attention control conditions will involve 2 components: face-to-face (individual) counseling sessions with a school nurse and an after-school (group) program. The intervention for the attention control group will not address physical activity. Both groups will respond to questionnaires at 0 (baseline) and 6 mos. Our "Girls on the Move" intervention is designed to help girls achieve physical activity recommendations (≥ 60 min. ≥ 5 days/wk.). The motivational, individually tailored counseling sessions with a school nurse and after-school physical activity club (3-5 times a wk. for 6 mos.) are designed to positively influence all cognitive and affective mediating variables of the Health Promotion Model.

SUMMARY:
Specific aims are:

1. Evaluate the feasibility of the intervention related to (1) girls' participation; (2) adherence to protocols; and (3) user and provider (nurse and PA Club instructors) satisfaction.
2. Explore if participants in the intervention group, compared to those in the control group, show improvement in the primary outcome of minutes of moderate to vigorous physical activity (MVPA; measured by accelerometer), and also secondary outcomes of self-report of MVPA, cardiovascular fitness, body mass index, percent body fat, and waist circumference at 6 months.
3. Explore if the primary outcome is mediated by cognitive (perceived benefits of PA, perceived barriers to PA,PA self-efficacy, social support, norms, models) and affective (enjoyment of PA) variables.
4. Explore if participants in the intervention group, compared to those in the control group, have greater minutes of MVPA at 7 months.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of and obtain preliminary evidence of efficacy for a 6-month "Girls on the Move" intervention (guided by the Health Promotion Model and Social Cognitive Theory). The intervention involves motivational, individually tailored counseling plus after-school physical activity (PA) to increase moderate to vigorous physical activity (MVPA) and cardiovascular (CV) fitness, as well as improve body composition and cognition and affective responses related to MVPA among 6th-grade girls. Specifically, it consists of a 90-minute after-school PA Club that includes MVPA and 6 one-on-one monthly motivational, individually tailored counseling sessions with a registered (school) nurse during the school day to support each girl's continued MVPA. Applying the motivational interviewing communication style, the school nurse will individually tailor the counseling based upon each girl's key responses gleaned from computerized questionnaires assessing cognitive and affective variables related to MVPA. One middle school will be randomly assigned to receive the intervention and another to serve as attention control.

ELIGIBILITY:
Inclusion Criteria:

(1) 6th-grade girls (ages 10-12) (7th-graders if needed; up to and including age 14) who report not meeting national MVPA recommendations; (2) available and willing to participate 6 mos.; and (3) able to read, understand, and speak English (e.g., school nurse checks that girl is reading at grade level or enrolled in remedial course).

Exclusion criteria:

(1) Involved in school or community sports or other organized PAs or lessons, such as dance, martial arts, gymnastics, or tennis, that involve MVPA and require participation 3 or more days/wk. during every season of the school year; and (2) a health condition limiting or precluding safe MVPA.

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate to vigorous physical activity | baseline and 6 months

SECONDARY OUTCOMES:
self-report of moderate to vigorous physical activity | baseline and 6 months
cardiovascular fitness | baseline and 6 months
Body mass index (BMI) | baseline and 6 months
percent body fat | baseline and 6 months
waist circumference | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine B Robbins, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

REFERENCES:
- [Result] Robbins LB, Pfeiffer KA, Maier KS, Lo YJ, Wesolek Ladrig SM. Pilot intervention to increase physical activity among sedentary urban middle school girls: a two-group pretest-posttest quasi-experimental design. J Sch Nurs. 2012 Aug;28(4):302-15. doi: 10.1177/1059840512438777. Epub 2012 Apr 3. PMID 22472632
- [Result] Robbins LB, Pfeiffer KA, Maier KS, Ladrig SM, Berg-Smith SM. Treatment fidelity of motivational interviewing delivered by a school nurse to increase girls' physical activity. J Sch Nurs. 2012 Feb;28(1):70-8. doi: 10.1177/1059840511424507. Epub 2011 Oct 4. PMID 21970862
- [Result] Vanden Bosch ML, Robbins LB, Pfeiffer KA, Kazanis AS, Maier KS. Demographic, cognitive, affective, and behavioral variables associated with overweight and obesity in low-active girls. J Pediatr Nurs. 2014 Nov-Dec;29(6):576-85. doi: 10.1016/j.pedn.2014.06.002. Epub 2014 Jun 17. PMID 25027734